CLINICAL TRIAL: NCT00214851
Title: The Use of Kineret (Anakinra) in the Treatment of Familial Cold Urticaria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Atlantic Provinces Dermatology Association (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDHA002
Record Dates: First submitted 2005-09-21; First posted 2005-09-22 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2008-05

CONDITIONS: Familial Cold Urticaria
Keywords: Familial Cold Urticaria; Kineret (anakinra); Interleukin 1 beta; C-Reactive Protein; Serum Amyloid A protein
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Kineret (anakinra) — Kineret (anakinra 100 mg. s/c daily x 4 weeks

SUMMARY:
An open labelled trial of Kineret (anakinra) induction therapy (100mg./day) in over a four week period in the treatment of Familial Cold Urticaria.

Familial Cold Urticaria (FCU) is a rare autosomal dominant condition manifesting symptoms triggered by exposure to cold and variable in expression. Currently there is no standard reliable agent available for the treatment of patients with FCU.This study will evaluate the efficacy of Kineret (anakinra), an interleukin 1 receptor antagonist in induction and maintenance therapy in patients with FCU.

DETAILED DESCRIPTION:
Product: Kineret (anakinra) Protocol title: The Use of Kineret (anakinra) in the Treatment of Familial Cold Urticaria (FCU) Target Disease: Familial Cold Urticaria Patients: 8 patients all previously diagnosed with FCU and living close to Moncton, N.B.

Study Objectives:

* To assess the efficacy of Kineret (anakinra) 100mg. given subcutaneously daily in subjects with FCU.
* To demonstrate the use of CRP and SAA as objective laboratory markers of the effectiveness of treatment.
* To determine the effect of Kineret (anakinra)on the quality of life of patients with FCU.

Study design: An open-labelled trial of Kineret (anakinra) induction therapy (100mg./day) over a four week period.

Treatment regimens: After initial clinical and laboratory assessment, the patients will receive Kineret (anakinra) 100mg. daily for four weeks. They will be observed for two further weeks without the medication.

Route of administration: Subcutaneous injection Interval between first and last dose of active study agent: 4 weeks Duration of study participation: 8 weeks Number of subjects: 8 Number of sites: 1 Interim analysis: Daily patient diary; weekly follow-up phone calls; CRP reports

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older at the time of enrollment; may be male or female
* Must be previously diagnosed with Familial Cold Urticaria (FCU)
* Must react with at least one of the symptoms of FCU in the summer months at least four times per week sufficiently to interfere with ordinary daily activities or inhibit normal life enjoyment.
* Women must be willing to have a pregnancy test and if necessary, use contraceptive measures.

Exclusion Criteria:

* Receiving any systemic medications/treatments that could affect FCU.
* Pregnancy, nursing or planning pregnancy, or, have recently been pregnant to less than three months development and with a history of serious birth defect.
* Have had any previous treatment with Kineret (anakinra) or any therapeutic agent targeted at IL-1 blockade.
* Have used any investigational drug within the previous 1 month or five times the half life of the investigational agent, whichever is longer, or 3 months for any biologic of unknown half life.
* Have received any systemic medication or treatments that could affect the symptoms of FCU such as antihistamines, corticosteroid drugs, NSAIDS, anabolic medications or Ketotifen within 2 weeks of the baseline visit.
* Have any known malignancy or have a history of malignancy within the previous five years (with the exception of basal or squamous cell carcinoma of the skin that has been treated with no evidence of recurrence).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2005-09; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of kineret (anakinra) 100mg./day in subjects with familial cold urticaria. | Eight weeks

SECONDARY OUTCOMES:
To demonstrate the use of C-Reactive Protein (CRP) and Serum Amyloid A Protein (SAA) levels as objective laboratory indicators of effective treatment and to compare the results of two different laboratory methods for the estimation of CRP | Eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Laura A. Finlayson MD FRCPC, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Queen Elizabeth Health Sciences Centre, Halifax, Nova Scotia, Canada